CLINICAL TRIAL: NCT05150496
Title: A Phase IIb Randomized Double-Blinded Positive Controlled Trial to Evaluate the Immunogenicity and Safety Study of the 3rd Booster Dose Using the High or Medium Dose of Inactivated (CoronaVac®) Vaccine in Healthy Adults Who Have Completed Two Doses of CoronaVac® or the mRNA Vaccine (Comirnaty) in Turkey
Brief Title: Immunogenicity and Safety Study of the 3rd Booster Dose Using the High or Medium Dose of Inactivated (CoronaVac®) Vaccine in Healthy Adults in Turkey
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: The plan has changed
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-nCOV-2002
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Two doses CoronaVac® + one dose medium-dose CoronaVac® (Experimental): 200 participants who were vaccinated with CoronaVac® will be given one dose booster immunization using medium-dose CoronaVac®3-8 months after their second dose
  Interventions: Biological: Medium-dose COVID-19 Vaccine(Vero Cell),Inactivated
- Two doses CoronaVac® + one dose high-dose CoronaVac® (Experimental): 200 participants who were vaccinated with CoronaVac® will be given one dose booster immunization using high-dose CoronaVac® 3-8 months after their second dose
  Interventions: Biological: High-dose COVID-19 Vaccine(Vero Cell),Inactivated
- Two doses Comirnaty + one dose medium-dose CoronaVac® (Experimental): 120 participants were vaccinated with Comirnaty will be given one dose booster immunization using medium-dose CoronaVac® 6-8 months after their second dose
  Interventions: Biological: Medium-dose COVID-19 Vaccine(Vero Cell),Inactivated
- Two doses Comirnaty + one dose high-dose CoronaVac® (Experimental): 120 participants were vaccinated with Comirnaty will be given one dose booster immunization using one dose high-dose CoronaVac® 6-8 months after their second dose
  Interventions: Biological: High-dose COVID-19 Vaccine(Vero Cell),Inactivated

INTERVENTIONS:
Biological: Medium-dose COVID-19 Vaccine(Vero Cell),Inactivated — Medium-dose COVID-19 Vaccine(Vero Cell),Inactivated: 600SU inactivated SARS-CoV-2 virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: Medium-dose CoronaVac®
  Arms: Two doses Comirnaty + one dose medium-dose CoronaVac®; Two doses CoronaVac® + one dose medium-dose CoronaVac®
Biological: High-dose COVID-19 Vaccine(Vero Cell),Inactivated — High-dose COVID-19 Vaccine(Vero Cell),Inactivated:1200SU inactivated SARS-CoV-2 virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: High-dose CoronaVac®
  Arms: Two doses Comirnaty + one dose high-dose CoronaVac®; Two doses CoronaVac® + one dose high-dose CoronaVac®

SUMMARY:
This is a randomized, double-blinded, and positive-controlled Phase IIb clinical trial of COVID-19 vaccine (CoronaVac®) manufactured by Sinovac Research & Development Co., Ltd.The purpose of this study is to evaluate the immunogenicity of using the high (1200SU) or medium (600SU) dose of CoronaVac® as the booster dose.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, and positive-controlled phaseⅡb clinical trial of 640 participants aged 18 years and above, who have completed 2 doses of inactivated COVID-19 vaccine (CoronaVac®) or mRNA COVID-19 vaccine (Comirnaty) as the primary vaccination. Participants will be enrolled and randomly assigned into two arms at a ratio of 1:1 to receive a booster dose of medium-dose (600SU) or high-dose (1200SU) COVID-19 Vaccine. For those who were vaccinated with CoronaVac®, the booster dose will be given 3-8 months after their second dose. For those who were vaccinated with Comirnaty, the booster dose will be given 6-8 months after their second dose. Each participant will be collected 5.0 ml blood sample before vaccination and 14 days,3 months and 6 months after booster immunization.Immunogenicity assessments will be determined by neutralizing antibodies in all participants.In addition,all participants will be monitored for immediate reactions (within 30 minutes) after the booster dose vaccination, adverse events of special interest (AESIs) and serious adverse events (SAEs) for 12 months after booster dose inoculation. In addition, all participants in will be monitored for local and systemic solicited adverse events (AEs) within 7 days and the unsolicited AEs within 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 years and above, who have received 2 prior doses of inactivated COVID-19 vaccine (CoronaVac®) or mRNA COVID-19 vaccine (Comirnaty), with the second dose given 3-8 months (for CoronaVac® recipients) and 6-8 months (for Comirnaty recipients) prior to the day of booster vaccination in the present study;
* Antigen rapid testing negative at the day of enrollment on site or with a PCR negative result within 72 hours before enrollment;
* The participants are able to understand and sign the informed consent voluntarily;
* Female participants who have a negative pregnancy test on the day of vaccination, and not currently breastfeeding;
* The participants are planning to be living in Turkey for the following 1 year after attending this study;
* The participants must be willing to provide verifiable identification (in accordance with the local regulations), has means to be contacted and to contact the investigator during the study.

Exclusion Criteria:

* History of confirmed or currently with the infection of SARS-CoV-2 prior to randomization;
* Any prior administration of another investigational coronavirus vaccine or current/planned simultaneous participation in another interventional study to prevent or treat COVID-19;
* Known allergy to vaccines or vaccine ingredients, and serious adverse reactions to vaccines, such as urticaria, dyspnea, angioneurotic edema;
* Serious chronic disease, serious cardiovascular disease, hypertension and diabetes that cannot be controlled by drugs, hepatorenal disease, malignant tumor, etc;
* Acute central nervous system diseases such as encephalitis/myelitis, acute disseminating encephalomyelitis, and related disorders;
* Receipt of blood/plasma products or immunoglobulins in the past 3 months before vaccination in this study;
* Participation in other studies involving study intervention within 30 days prior to vaccination in this study;
* Receipt of attenuated live vaccines in the past 14 days prior to vaccination in this study;
* Receipt of inactivated or subunit vaccines in the past 7 days prior to vaccination in this study;
* Acute exacerbation or presentation of stable chronic diseases (including but not limited to asthma, migraine, gastrointestinal disorder, etc.);
* Acute febrile illness with axillary temperature >37.5°C on the day of vaccination; enrollment could be considered if the fever is absent for 72 hours prior to vaccination;
* According to the investigator's judgment, the participant has any other factors that might interfere with the results of the clinical trial or pose additional risk to the participant due to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity index-GMT of neutralizing antibodies | 14 days (14-28 days) after the booster dose vaccination
  GMT of neutralizing antibodies on 14 days (14-28 days) after the booster dose vaccination

SECONDARY OUTCOMES:
Immunogenicity index-Seropositivity rate of neutralizing antibodies | 14 days (14-28 days) after the booster dose vaccination
  Seropositivity rate of neutralizing antibodies on 14 days (14-28 days) after the booster dose vaccination
Immunogenicity index-GMI of neutralizing antibodies | 14 days (14-28 days) after the booster dose vaccination
  GMI of neutralizing antibodies on 14 days (14-28 days) after the booster dose vaccination
Immunogenicity index-The seropositivity rate of neutralizing antibody | At 3 (±2 weeks) and 6 (±2 weeks) months after the booster dose vaccination
  Seropositivity rate of neutralizing antibody at 3 (±2 weeks) and 6 (±2 weeks) months after the booster dose vaccination
Immunogenicity index-GMT of neutralizing antibody | At 3 (±2 weeks) and 6 (±2 weeks) months after the booster dose vaccination
  GMT of neutralizing antibody at 3 (±2 weeks) and 6 (±2 weeks) months after the booster dose vaccination
Safety index-Occurrence, intensity, duration, and relationship of solicited local and systemic AEs | 7 days following the booster dose vaccination
  Occurrence, intensity, duration, and relationship of solicited local and systemic AEs for 7 days following the booster dose vaccination
Safety index-Occurrence, intensity, duration, and relationship of unsolicited AEs | 28 days post booster vaccination
  Occurrence, intensity, duration, and relationship of unsolicited AEs for 28 days post booster vaccination
Safety index-Occurrence and relationship of SAEs | From the booster dose to 12 months post booster vaccination
  Occurrence and relationship of SAEs (from the booster dose to 12 months post booster vaccination)
Safety index-Occurrence and relationship of AESI | From the booster dose to 12 months post booster vaccination
  Occurrence and relationship of AESI (from the booster dose to 12 months post booster vaccination)

OTHER OUTCOMES:
Immunogenicity index-The seropositivity rate of neutralizing antibodies | Before vaccination, 14 days (14-28 days) , 3-month (±2 weeks), and 6-month (±2 weeks) after the booster dose vaccination
  The seropositivity rate of neutralizing antibodies before vaccination, 14 days (14-28 days) , 3-month (±2 weeks), and 6-month (±2 weeks) after the booster dose vaccination
Immunogenicity index-GMT of neutralizing antibodies | Before vaccination, 14 days (14-28 days) , 3-month (±2 weeks), and 6-month (±2 weeks) after the booster dose vaccination
  GMT of neutralizing antibodies before vaccination, 14 days (14-28 days) , 3-month (±2 weeks), and 6-month (±2 weeks) after the booster dose vaccination
Immunogenicity index-GMI of neutralizing antibodies | Before vaccination, 14 days (14-28 days) , 3-month (±2 weeks), and 6-month (±2 weeks) after the booster dose vaccination
  GMI of neutralizing antibodies before vaccination, 14 days (14-28 days) , 3-month (±2 weeks), and 6-month (±2 weeks) after the booster dose vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Enes Seyda Şahiner, Doctor, Principal Investigator — Republic of Turkey Ministry of Health Ankara City Hospital Department of Internal Diseases
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University Faculty of Medicine, Department of Internal Diseases / Infectious Diseases and Clinical Microbiology Unit, Ankara
  - Republic of Turkey Ministry of Health Ankara City Hospital Department of Internal Diseases, Ankara